CLINICAL TRIAL: NCT03389243
Title: Influence of SPI-guided Analgesia With Preemptive Analgesia Using Either Paracetamol or Metamizole on the Presence of Oculocardiac Reflex, Postoperative Pain, Postoperative Nausea and Vomiting in Patients Undergoing VRS Under General Anaesthesia: a Randomised, Controlled Trial
Brief Title: Paracetamol and Metamizole With SPI-guided Anaesthesia for VRS
Acronym: P&MSPIVRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Collaborators: Silesian University of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: SilesianMUKOAiIT7
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2022-01

CONDITIONS: Vitreoretinal Surgeries; Postoperative Nausea and Vomiting; Postoperative Pain
Keywords: Surgical Pleth Index (SPI); General Anaesthesia (GA),; Numerical Rating Scale (NRS); Adequacy of Anaesthesia (AoA); Oculocardiac reflex (OCR); paracetamol; metamizole
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Dipyrone; Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- metamizol (Experimental): analgesic drug
  Interventions: Drug: paracetamol; Drug: paracetamol and metamizole
- paracetamol (Experimental): analgesic drug
  Interventions: Drug: Metamizol; Drug: paracetamol and metamizole
- metamizole & paracetamol (Experimental): analgesic drugs
  Interventions: Drug: Metamizol; Drug: paracetamol

INTERVENTIONS:
Drug: Metamizol — in group M patients will receive pre-emptive analgesia using intravenous infusion of metamizol in a single dose of 1,25 gram
  Other Names: Pyralgin
  Arms: metamizole & paracetamol; paracetamol
Drug: paracetamol — in group P patients will receive pre-emptive analgesia using intravenous infusion of metamizol in a single dose of 1,25 gram
  Arms: metamizol; metamizole & paracetamol
Drug: paracetamol and metamizole — in group PM patients will receive pre-emptive analgesia using intravenous infusion of metamizol in a single dose of 1,25 gram and paracetamol in a dose of 1 gram
  Arms: metamizol; paracetamol

SUMMARY:
The aim of this randomized trial is to assess the efficacy of preemptive analgesia using paracetamol or metamizole or both of them under SPI-guided anaesthesia for vitreoretinal surgery (VRS), presence of PONV (postoperative nausea and vomiting) and oculocardiac reflex (OCR) and compare Numerical Rating Scale (NRS) with Surgical Pleth Index (SPI) for monitoring pain perception postoperatively.

Patients will receive general anaesthesia combined with either preemptive analgesia using preemptive intravenous infusion of 1,0 g of metamizol or preemptive intravenous infusion of 1,0 g of acetaminophen or both of them together.

DETAILED DESCRIPTION:
Monitoring depth of anaesthesia using spectral entropy (SE) and quality of neuromuscular block are routine in modern anaesthesia, whereas monitoring of analgesia still requires further studies. Recently, the Surgical Pleth Index (SPI) was added as a surrogate variable showing the nociception-antinociception balance into abovementioned parameters constituting a novel approach in monitoring patients intraoperatively, known as adequacy of anaesthesia (AoA) or tailor-made anaesthesia.

Different options of preemptive analgesia are used to decrease the postoperative pain perception as well as diminish the rate of PONV by deceasing intraoperative consumption of intravenous narcotic analgesics

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate in the study
* written consent to undergo general anaesthesia alone or combined with different techniques of pre-emptive analgesia and vitreoretinal surgery

Exclusion Criteria:

* history of allergy to local paracetamol or metamizole
* necessity of administration of vasoactive drugs influencing SPI monitoring
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
pain perception intraoperatively | intraoperatively
  The investigators will compare the efficacy of analgesia intraoperatively according to used preoperatively intravenous infusions . The investigators will administer a rescue dose of fentanyl intravenously in a dose of 1 mcg per kg of body weight in the case when SPI value increases over 10 points in SPI scale every 5 minutes until SPI value decreases back to baseline value. Additionally, the investigators will analyse rescue fentanyl consumption in abovementioned groups

SECONDARY OUTCOMES:
pain perception postoperatively | up to one hour after discharge to postoperative unit.
  The investigators will compare the efficacy of analgesia postoperatively according to technique of analgesia used preoperatively: intravenous infusion of either metamizol or paracetamol or both of them. The investigators use NRS and compare it with SPI values.
PONV | up to 24 hours
  The investigators will compare the presence of PONV after emergence from GA in studied groups. The investigators will observe patients postoperatively and record any incidence of nausea or vomiting and in the abovementioned case the investigators will administer a standard dose of antiemetic drug.
oculocardiac reflex rate | intraoperatively
  The investigators will compare the rate of presence of OCR intraoperatively in studied groups

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Silesia, Sosnowiec, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
article in Pharmaceuticals in 2024, case reports
Supporting Information: ICF
Time Frame: three years

REFERENCES:
- [Result] Gruenewald M, Herz J, Schoenherr T, Thee C, Steinfath M, Bein B. Measurement of the nociceptive balance by Analgesia Nociception Index and Surgical Pleth Index during sevoflurane-remifentanil anesthesia. Minerva Anestesiol. 2015 May;81(5):480-9. Epub 2014 Jul 17. PMID 25032676
- [Result] Gruenewald M, Ilies C, Herz J, Schoenherr T, Fudickar A, Hocker J, Bein B. Influence of nociceptive stimulation on analgesia nociception index (ANI) during propofol-remifentanil anaesthesia. Br J Anaesth. 2013 Jun;110(6):1024-30. doi: 10.1093/bja/aet019. Epub 2013 Mar 6. PMID 23471754
- [Result] Gruenewald M, Ilies C. Monitoring the nociception-anti-nociception balance. Best Pract Res Clin Anaesthesiol. 2013 Jun;27(2):235-47. doi: 10.1016/j.bpa.2013.06.007. PMID 24012235
- [Result] Gruenewald M, Willms S, Broch O, Kott M, Steinfath M, Bein B. Sufentanil administration guided by surgical pleth index vs standard practice during sevoflurane anaesthesia: a randomized controlled pilot study. Br J Anaesth. 2014 May;112(5):898-905. doi: 10.1093/bja/aet485. Epub 2014 Feb 16. PMID 24535604
- [Result] Fekrat S, Elsing SH, Raja SC, Campochiaro PA, de Juan E Jr, Haller JA. Eye pain after vitreoretinal surgery: a prospective study of 185 patients. Retina. 2001;21(6):627-32. doi: 10.1097/00006982-200112000-00010. PMID 11756886
- [Result] Mandelcorn M, Taback N, Mandelcorn E, Ananthanarayan C. Risk factors for pain and nausea following retinal and vitreous surgery under conscious sedation. Can J Ophthalmol. 1999 Aug;34(5):281-5. PMID 10486687